CLINICAL TRIAL: NCT02845765
Title: Evaluation of Vascularization of the Fundus Oculi in Patients With Erectile Dysfunction as Barometer of Patient's Health
Brief Title: Fundus Oculi and Erectile Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Querques Giuseppe, Head-Medical retina & Imaging unit, Ospedale San Raffaele
Other Study IDs: N.2015 FundusOculi_DE
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2019-07

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; ED; Fundus Oculi; Retinal Vascularization; International Index of Erectile Function Questionnaire; IIEF; Dynamic Vessel Analyzer; DVA; Phosphodiesterase type 5 Inhibitor; PDE5Is
MeSH Terms: conditions — Erectile Dysfunction | interventions — Phosphodiesterase 5 Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with erectile dysfunction: Patients with erectile dysfunction characterized by the inability to develop or maintain an erection of the penis during sexual activity. Patients will be examined with Dynamic Vessel Analyzer (DVA) at baseline and 6 months after therapy with Phosphodiesterase type 5 Inhibitor (PDE5I).
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Drug: Phosphodiesterase type 5 Inhibitor (PDE5I)
- Subject healthy volunteers: Patients without erectile dysfunction or ocular disease. Patients will be examined with Dynamic Vessel Analyzer (DVA) at baseline
  Interventions: Device: Dynamic Vessel Analyzer (DVA)

INTERVENTIONS:
Device: Dynamic Vessel Analyzer (DVA)
Drug: Phosphodiesterase type 5 Inhibitor (PDE5I)
  Groups: Patients with erectile dysfunction

SUMMARY:
The purpose of this study is to evaluate the correlation between fundus oculi's vascularization in patients with erectile dysfunction and not, and, in the same patients, before and after using drugs for ED.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the correlation between fundus oculi's vascularization in patients with erectile dysfunction and not, and, in the same patients, before and after using drugs for ED.

In this monocentric, prospective, observational case-control study 40 eyes of 40 patients affected by erectile dysfunction and 20 healthy age-matched controls will be enrolled.

Patients will undergo DVA examination at baseline and 6 months after PDE5I therapy. Healthy subjects will be examined with DVA at baseline only.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with erectile dysfunction diagnosis (organic and psychogenic);
* Subjects with Erectile Dysfunction diagnosis defined by IIEF score ≤ 25
* Subjects with stable partner for at least 6 months and sexually active.
* Subjects aged between 40 - 60 years;
* Signature of informed consent for patients

Exclusion Criteria:

* Subjects with ED secondary diagnosis to hormonal alterations (i.e. hypogonadism, hypo / hyperthyroidism, hyperprolactinemia);
* Subjects with a diagnosis of ED post-traumatic and iatrogenic, since after pelvic surgery;
* Subjects suffering from any ocular pathology that involves use of contact lenses and / or glasses;
* Subjects smoking;
* Individuals with uncontrolled systemic diseases;
* All persons who do not confirm at least one criterion for inclusion.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * n. 40 patients with erectile dysfunction haracterized by the inability to develop or maintain an erection of the penis during sexual activity
  * n. 20 subject healthy volunteers without erectile dysfunction or ocular desease
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Static and dynamic retinal vessels diameter | Baseline and after 6 month of therapy
  Analysis of the presence and prevalence of retinal vascularization alterations using Dynamic Vessel Analyzer (DVA) in patients with Erectile Dysfunction and in subject healthy volunteers.

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) Questionnaire | After 6 month of therapy
  Revaluation of the correlation between Erectile Dysfunction and Fundus Oculi vascularization after 6 month of therapy for ED.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, PhD, Principal Investigator — University Vita-Salute, San Raffaele Hospital - Milan
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided